CLINICAL TRIAL: NCT04571697
Title: Comparing Rates of Dementia and Alzheimer's Disease in Patients Initiating Methotrexate Versus Those Initiating Anti-TNF-α Therapy
Brief Title: A Study of Comparing Rates of Dementia and Alzheimer's Disease in Participants Initiating Methotrexate Versus Those Initiating Anti-tumor Necrosis Factor (TNF)-Alpha Therapy
Status: Completed | Type: Observational
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: CR108890; PCSNSP002938 (Other: Janssen Research & Development, LLC)
Record Dates: First submitted 2020-09-25; First posted 2020-10-01 (Actual); Last update posted 2025-04-27 (Actual); Status verified 2025-04

CONDITIONS: Dementia; Alzheimer Disease
MeSH Terms: conditions — Dementia; Alzheimer Disease | interventions — Methotrexate

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes

GROUPS / COHORTS (1):
- Participants Initiating Therapy with Methotrexate or Anti-TNF: Data will be collected for participants initiating therapy with either methotrexate or an anti-tumor necrosis factor (TNF) from united states (US) claims databases: optum de-identified clinformatics data mart database and IBM marketscan medicare supplemental database (MDCR). Data collection period: 01-Jan-2000 through 31-Jul2019.
  Interventions: Drug: Methotrexate; Drug: Anti-TNF

INTERVENTIONS:
Drug: Methotrexate — No intervention or treatment will be administered as part of this study. Data of participants with first claim for a methotrexate in the patient's history are included.
Drug: Anti-TNF — No intervention or treatment will be administered as part of this study. Data of participants with first claim for an anti-TNF in the patient's history are included. Anti-TNF includes infliximab, golimumab, etanercept, certolizumab, and adalimumab.

SUMMARY:
The purpose of the study is to compare the risk of dementia in participants diagnosed with rheumatoid arthritis (RA) exposed to anti-tumor necrosis factor (TNF) therapy versus those exposed to methotrexate.

ELIGIBILITY:
Inclusion Criteria:

* At least one claim for methotrexate or anti-TNF therapy during the study period. First medication received is the index medication, and date of first receipt is the index date
* 365 days of continuous pre-index observation immediately prior to the index date
* Participants have at least two occurrences of a diagnosis of rheumatoid arthritis within 365 days before and including the index date
* No prior use of methotrexate or an anti- tumor necrosis factor (TNF) therapy at any time prior to the index date
* Cohort follow-up persists until end of continuous observation or filling the comparator drug

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Study population consists of participants who are new user of Anti-TNF therapy diagnosed with dementia and alzheimer's disease.
Sampling Method: Non-Probability Sample
Enrollment: 34647 (Actual)
Dates: Start 2020-09-28 (Actual); Primary Completion 2020-10-27 (Actual); Study Completion 2020-10-27 (Actual)

PRIMARY OUTCOMES:
Newly Diagnosed Dementia Cases | 365 days
  An outcome of dementia requires at least two diagnosis codes international classification of diseases, ninth revision, clinical modification (ICD-9-CM) or international classification of diseases, tenth revision, clinical modification (ICD-10-CM) for dementia within 365 days of each other.

SECONDARY OUTCOMES:
Newly Diagnosed Alzheimer's Disease (AD) Cases | 365 days
  An outcome of AD requires at least two diagnosis codes (ICD-9-CM or ICD-10-CM) for AD within 365 days of each other.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (1):
- Janssen R&D, Titusville, New Jersey, United States